CLINICAL TRIAL: NCT04085926
Title: Sealed Therapeutic Shoe vs. Total Contact Cast as Treatment of Diabetic Foot Ulcers: a Multicenter RCT
Brief Title: Sealed Therapeutic Shoe as Treatment of Diabetic Foot Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with recruting participants
Sponsor: Region Örebro County (Other)
Collaborators: Forte (Industry)
Responsible Party: Principal Investigator, Gustav Jarl, Associate Professor, Certified Prosthetist and Orthotist, Region Örebro County
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18RS6667
Record Dates: First submitted 2019-09-02; First posted 2019-09-11 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Foot
Keywords: Wound Healing; Casts, Surgical; Shoes
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The primary outcome (ulcer healing) will be assessed by a cast technician not blinded to group allocation, but it will be verified from a photograph by a blinded assessor. The statistician comparing the primary outcome between groups will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sealed shoe (Experimental): Therapeutic footwear including off-the-shelf therapeutic shoes and custom-made insoles. The shoe on the ulcerated foot is "sealed", i.e., made irremovable, with a plastic band.
  Interventions: Device: Sealed therapeutic shoe
- Total contact cast (Active Comparator): A irremovable custom-made total Contact cast enclosing the foot and shin
  Interventions: Device: Total contact cast

INTERVENTIONS:
Device: Sealed therapeutic shoe — Off-the-shelf therapeutic shoe and custom-made insole
  Arms: Sealed shoe
Device: Total contact cast — Custom-made total contact cast
  Arms: Total contact cast

SUMMARY:
Total contact casts (TCCs) are effective treatment of plantar diabetic foot ulcers because they effectively offload the ulcer and are non-removable, resulting in high adherence to using the device. However, TCCs are not widely used in clinical practice because they negatively impact gait and daily activities. A new treatment concept was invented, sealed therapeutic shoe, where a shoe with a custom-made insole offloads the ulcer, and the shoe is rendered irremovable to be worn day and night, like a TCC.

In this multicenter randomized controlled trial (RCT), 150 participants will be recruited and randomized to two treatment arms: TCC or sealed therapeutic shoe. The primary outcome is ulcer healing, secondary outcomes include (but are not limited to) skin complications, glycemic control, body mass index, gait function, balance, quality of life, physical activity, and health economics.

DETAILED DESCRIPTION:
Data for the primary outcome of 112 participants are needed but the aim is to recruit 150, if possible within a reasonable time frame, to take drop-out into account.

Participants are randomized (blocked randomization, stratified for ulcer site and study center) to either treatment with a sealed therapeutic shoe or total contact cast.

Each participant will be assessed by a cast technician during the treatment period (for ulcer healing and skin complications) and be assessed by a physiotherapist on five occasions: at baseline, approximately 4 weeks into treatment and 1, 6 and 12 months after treatment end. On these occasions the physiotherapist will perform different tests (gait, balance, ankle strength and flexibility, bone mass density in heel bone, etc) and participants will answer questionnaires and have their physical activity measured for 7 days with an activity monitor.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with diabetes mellitus (any kind)
* Foot ulcer under metatarsal heads

Exclusion Criteria:

* large ulcer (3-5 metatarsal heads)
* critical ischemia (defined as toe pressure <30 mmHg or TcPO2 <30 mmHg)
* uncontrolled infection (IWGDF infection grade 4, or grade 3 if not treatment against infection has been administered)
* Active Charcot foot
* foot deformities that necessitate custom-made shoes
* inability to speak/read Swedish.
* People with increased risk that side-effects will not be discovered or reported (dementia, abuse of alcohol or drugs, intellectual disability, etc.) if the person do not have appropriate social support, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with healed foot ulcers at 12 weeks | 12 weeks after treatment is initiated
  Defined as complete epithelization, verified on a second occasion at least 14 days later. Primary outcome measure is proportion of ulcers healed in each Group after 12 weeks of treatment.

SECONDARY OUTCOMES:
Number of participants with skin complications through study completion (treatment period, on average 12 weeks) | Through study completion (treatment period, on average 12 weeks)
  abrasions, iatrogenic ulcers, blisters, etc.
Average level of plasma glucose concentration, measured as glycated haemoglobin (HbA1c) | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  Blood sample of HbA1c
Body mass index | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  weight (kg) divided by squared length (m)
Gait function assessed with 10 m Walk test, mean value | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  Time to complete test, longer time is worse
Gait function assessed with Timed up and go test, mean value | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  Time to complete test, longer time is worse
Mean score on Berg balance scale | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  Total sum score is used, range 0-56 (higher is better)
Calf muscle atrophy measured as maximal calf circumference | Baseline, 1, 6, and 12 months after treatment end
  Average values (cm) are reported
General quality of Life measured with Short form 36 (SF-36) | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  Mean values, score range 0-100 (higher is better)
General quality of Life measured with Euroqol 5 dimension 5 levels (EQ-5D-5L) | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  Mean values, score range 0-1 (higher is better)
Disease-specific quality of life measured with Diabetic foot ulcer scale -short form | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  Mean values, score range 29-145 (lower is better)
Mean daily number of steps measured with ActivPAL activity monitor | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  Mean daily number of steps measured with ActivPAL activity monitor
Mean daily time spent sitting measured with ActivPAL activity monitor | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  Mean daily time spent sitting measured with ActivPAL activity monitor
Mean daily time spent laying measured with ActivPAL activity monitor | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  Mean daily time spent laying measured with ActivPAL activity monitor
Mean daily time spent standing measured with ActivPAL activity monitor | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  Mean daily time spent standing measured with ActivPAL activity monitor
Physical activity measured with the Swedish National Board of Health and Welfare's indicator questions | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  3 items (intense activity, moderate activity, sitting time), each with 7 response alternatives (higher score is better)
Bone mass density in heel bone | Baseline, 1, 6, and 12 months after treatment end
  Dual-energy X-ray absorptiometry (DXA) of calcaneus
Internal locus of control measured with two items from Form C of the Multidimensional Health Locus of Control (MHLC-C) scale | Baseline, approx. 4 weeks into treatment, 1, 6, and 12 months after treatment end
  2 items, analyzed separately, score range 1-5 per item (lower is better)
Ankle range of motion (dorsal flexion) | Baseline, 1, 6, and 12 months after treatment end
  goniometer, standardized measurement method
Ankle strength (plantar and dorsal flexion) | Baseline, 1, 6, and 12 months after treatment end
  dynamometer, standardized measurement method
Adherence to using therapeutic footwear assessed with 2 self-report questions adapted from the Questionnaire for persons with a transfemoral amputation | Baseline, 1, 6, and 12 months after treatment end
  The 2 questions assess using time: number of days/week (range 0-7) and number of hours/day (6 categories). Higher score is better.
Satisfaction with treatment measured with visual analogue scale | approx. 4 weeks into treatment and 1 month after treatment
  Score range 0-100 (higher is better)
Number of new foot complications per study group after healing assessed with study-specific questionnaire and patient files | 6 and 12 months after treatment end
  Foot complications include new ulcers, Charcot foot, amputation, etc.
Out-patient health care consumption per participant assessed with study-specific questionnaire and patient files | 1, 6 and 12 months after treatment end
  Study-specific questionnaire with 5 items assessing number of visits (6 response categories, higher is worse) for 5 types of out-patient visits related to the foot ulcer. Patient files will also be used to assess the same variables.
In-patient health care consumption per participant assessed with study-specific questionnaire and patient files | 1, 6 and 12 months after treatment end
  Study-specific questionnaire where participants fill in each hospital admission (and time period) related to the foot ulcer. Also patient files will be used to assess the same variables.
Sick-leave from work (number of days per participant) during treatment period (average 12 weeks) and during the period after treatment end up to 12 months later, assessed with study-specific questionnaire and Swedish Social Insurance Agency's system data | 1, 6 and 12 months after treatment end
  Data from self-report questionnaire and Swedish Social Insurance Agency's system to assess number of days on sick leave

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Jarl, PhD, Principal Investigator — University Health Care Research Center, Region Örebro county
Locations (3):
- Sweden (3):
  - Mölndahls sjukhus, Gothenburg
  - Skånes Universitetssjukhus, Malmö, Malmo
  - Örebro Universitetssjukhus, Örebro

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT04085926/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT04085926/SAP_001.pdf